CLINICAL TRIAL: NCT06568120
Title: Effect of Using a Dragon Design Nebulizer Mask on Treatment Duration, Compliance and Fear in Children Presenting to the Emergency Department: A Randomized Controlled Trial
Brief Title: Effect of Using a Dragon Design Nebulizer Mask on Treatment Duration, Compliance and Fear in Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Koç University (Other)
Responsible Party: Principal Investigator, Eysan Hanzade Umac, Teaching and Research Assistant, Koç University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: kocuniversty
Record Dates: First submitted 2024-08-14; First posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Fear
Keywords: children; emergency room; fear
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Intervention Model Description: Randomized controlled study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (No Intervention): Children aged 3-6 who require nebulizer treatment in the emergency department, along with their families, will first be informed by one of the researchers. Then, children who are randomly assigned to the control group will be treated according to the institution's standard care procedures. The child and their family will be informed immediately before the treatment procedure. During the treatment, the child will be treated using a standard nebulizer mask appropriate for their age, in accordance with the institution's routine care procedures, and the parent will remain with the child throughout the treatment. The child's level of fear will be assessed by both the child and the nurse before and during the treatment. Additionally, the nurse will record the total duration of inhaler treatment and the child's adherence to the treatment.
- Dragon Mask Group (Experimental): Children who present to the emergency department and require nebulizer treatment will be randomly assigned to either the experimental or control groups. First, one of the researchers will meet with the child and their parent to provide information about the study. If the child and family agree to participate and are assigned to the experimental group, the child will be asked which mask design they prefer to use during the inhaler treatment: a dragon or a turtle. Additionally, before the treatment, the fear level of each child will be assessed by both the child and the nurse. During the treatment process, the children will receive nebulizer treatment appropriate for their age, and the duration and adherence to the treatment will be recorded by the nurse. Similarly, fear levels will be measured immediately before and during the treatment.
  Interventions: Device: dragon themed nebulizer masks

INTERVENTIONS:
Device: dragon themed nebulizer masks — This study is an experimental investigation aiming to evaluate the effect of a dragon-themed nebulizer mask (Figure 1), identified during a literature review by the researchers, on the duration of inhaler treatment application, treatment adherence, and children's fear levels. The dragon-designed nebulizer mask, with its colorful and toy-like appearance, is intended to calm children using pediatric aerosol masks. The mask is made of very soft, latex-free plastic, ensuring comfortable use for pediatric patients. It is compatible with all nebulizers and suitable for use in hospital settings. Unlike standard nebulizer masks, its appearance is designed with a dragon character specifically for pediatric patients. The mask is manufactured in China.
  Arms: Dragon Mask Group

SUMMARY:
Incorporating playful elements into medical devices has been shown to enhance the overall experience for pediatric patients. Children want a healthcare setting that is spacious, creative, imaginative, and contemporary. Additionally, a current retrospective study of 127,368 pediatric patients indicates that 71.26% of the visits involved children under five years old, and 23.64% of the cases were due to respiratory infections. This information highlights the prevalence of inhaler therapy in emergency departments, particularly among young children with respiratory issues. This study aims to evaluate the impact of using dragon/turtle-themed nebulizer masks on treatment application time, treatment adherence, and fear levels in children who present to emergency rooms. By addressing these environmental and procedural challenges, the study seeks to improve the overall experience and outcomes for pediatric patients undergoing inhaler therapy.

DETAILED DESCRIPTION:
The meaning of a disease or medical procedure may vary depending on the child's developmental milestones. Children aged 3-6 years, who are in the preoperational stage of cognitive development as defined by Piaget, often perceive hospital environments with curiosity and fear. This age group is characterized by a vivid imagination and limited understanding of the cause-and-effect relationship, which can lead to misconceptions about medical procedures and devices. For example, they may believe that they are being punished or that procedures or medical devices are more painful than they are. They may react with heightened anxiety, clinginess, or aggression. Even using face masks for aerosol therapy may cause distress in young children, as the masks can be perceived as scary or uncomfortable. Young children prefer a hospital environment that is bright, cheerful, warm, colorful, and comfortable. These environmental factors help reduce anxiety and create a more welcoming and less intimidating atmosphere for young patients.

Emergency rooms are often not designed to accommodate agitated young patients, featuring physical layouts that are not conducive to their care, noisy and chaotic environments, and limited access to therapeutic spaces. The care team may also lack the resources to manage agitated children effectively. On the other hand, recent studies have highlighted the importance of creating child-friendly medical environments to reduce anxiety and improve cooperation during treatment. This study aims to evaluate the impact of using dragon/turtle-themed nebulizer masks on treatment application time, treatment adherence, and fear levels in children who present to emergency rooms.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 3-6 years,
* Presenting to the emergency department with a respiratory problem (such as an upper respiratory tract infection) requiring nebulizer treatment,
* In general good health and suitable for nebulizer treatment (i.e., not having conditions like severe allergies or chronic respiratory failure),
* Possessing age-appropriate language and communication skills,
* Not previously familiar with the dragon-themed masks,
* Having parental consent.

Exclusion Criteria:

* Children with major medical or psychiatric comorbidities as reported by the physician, nurse, or parent,
* Children with a chronic health condition requiring regular nebulizer use (such as asthma),
* Children with a fever of 38°C (100.4°F) or higher,
* Children who have started treatment with sedative or anticonvulsant medications,
* Children and parents with visual, auditory, verbal, or cognitive impairments that would interfere with the use of the intervention equipment.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Fear - Child Fear Scale | Immediately before (baseline) treatment (approximately 5 minutes before), each child's fear level will be assessed by the child and the nurse. Similarly, fear levels will be measured again during the intervention.
  Thurillet et al. (2022) is used to learn about children's fears based on the autobiographical stories of children aged 4-12. The Turkish adaptation was made by Tavşan et al. in 2023. The scale consists of six facial expressions. The scale is graded with a score between 0 and 10 (graded gradually by two) along with fear and pain rating rates. It is seen that the first facial expression does not indicate fear, fear increases from right to left, and fear is most common in people's facial expressions.

SECONDARY OUTCOMES:
Duration of Treatment and Compliance | During the intervention, children will be given nebulizer treatment appropriate to their age, and the duration of treatment and compliance will be recorded by the nurse. This takes an average of 15-20 minutes.
  The start and end times of the inhaler treatment of the children in the experimental and control groups, as well as whether the children have complied with the treatment, will be evaluated with a form. The children in the experimental and control groups will be observed by nurses throughout the treatment period. The treatment durations of the children and their behaviors towards the treatment will be recorded as follows.

CONTACTS AND LOCATIONS:
Overall Officials: Eyşan Hanzade Savaş, PhD, Principal Investigator — Koç University
Locations (1):
- Koc University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No